CLINICAL TRIAL: NCT05211765
Title: Association of Respiratory Variation of Superior Vena Cava in Transthoracic View and Fluid Responsiveness in Critically Ill Patients
Brief Title: Respiratory Variation of Superior Vena Cava in Transthoracic View as a Fluid Responsiveness Predictor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Diego Ugalde Castillo, Assistant professor, University of Chile
Other Study IDs: 78/20
Record Dates: First submitted 2021-12-28; First posted 2022-01-27 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Superior vena cava transthoracic evaluation — The superior vena cava will be observed with a cardiac ultrasound machine, its diameter in different respiratory phases evaluated and compared with fluid response.

SUMMARY:
Fluid evaluation is relevant in critical care. Cardiac ultrasound is the first line of evaluation in hemodynamic characterization of patients in shock, to tailor therapy.

Fluid responsiveness predictors allow to better decide when to administer fluids, and transesophagic view of superior vena cava is an effective one. Recently a transthoracic view of the superior vena cava has been described.

The investigators aim to evaluate if the variations of superior vena cava can predict fluid responsiveness in critically il, ventilated patients.

Hypothesis: Respiratory variations of superior vena cava diameter, evaluated with transthoracic ultrasound, can predict fluid responsiveness

DETAILED DESCRIPTION:
Prospective evaluation of diameter variability of the superior vena cava by transthoracic echocardiography as fluid responsiveness predictor in critically ill patients:

Background Fluid administration is frequent in critically ill patients, particularly during reanimation and its empirical use is recommended as an initial step during this phase.

However, even though excess fluid administration is associated to negative outcomes fluid use is still being empirical and with scarce application of responsiveness predictors before its indication.

Different measurements or maneuvers exist, that allow clinicians to predict if a patient would present a positive fluid response, usually defined as cardiac output increasing 15% when infusing 500ml of crystalloids, and application of these predictive parameters could have clinical benefits on outcomes by avoiding inappropriate fluid administration.

As for the variables used, different types stand out. In general, flow or pressure variations originated in cardiothoracic interaction, auto-infusion and reduced fluid test evaluations such as the "mini" o "micro" fluid tests, in addition venous diameter variations in ultrasound evaluation with variable accuracy depending on the context. However, cardiothoracic interaction variables might have false positive results when right ventricular failure is present, given the cyclic increment on its afterload induced by positive pressure ventilation, reducing right ventricle stroke volume limiting its application in established or unknown and probable right heart failure if and advanced hemodynamic monitoring has not been performed to rule it out.

In this context, venous evaluations and reduced volume fluid test have advantages, and particularly in patients in shock under positive pressure ventilation, superior vena cava variation, being a better predictor than inferior vena cava. However, traditionally, superior vena cava can only be observed with transesophageal echocardiography and that can be a limitation in resource limited settings. Recently a new transthoracic acoustic window has been described, using a vertical left parasternal approach that allows evaluation of the superior vena cave, and initially, this approach shows a good correlation with the transesophageal measurement, and acceptable feasibility in the pilot study patients.

In this way, it can be postulated as possible, to evaluate if the variability of superior vena cava diameter on a transthoracic approach can be used as a fluid responsiveness predictor in critically ill patients on positive pressure ventilation.

Hypothesis Superior vena cava diameter respiratory variation evaluated with transthoracic ultrasound can predict fluid responsiveness in critically ill patients in positive pressure ventilation.

Objective To evaluate if superior vena cava respiratory diameter variation is associated with fluid responsiveness, when compared with the mini fluid infusion of 100ml evaluated with expiratory left ventricle outflow tract velocity time integral (LVOT-VTI) before and after fluid administration.

Methods

After evaluation, inclusion and exclusion criteria checking:

A basal echocardiography is performed, main pattern and clinical data are recorded (age, sex, weight, height, main diagnosis, secondary diagnosis, length of stay, surgical procedures, sequential organ failure assesment (SOFA) score, renal replacement therapy), respiratory (ventilator mode, tidal volume, respiratory rate, positive end expiratory pressure (PEEP), plateau pressure, peak inspiratory pressure, autoPEEP, fraction of inspired oxygen (FiO2), I:E relation, total inspiratory time), hemodynamic data from unit monitors. (cardiac rate, systolic pressure, diastolic pressure, mean pressure, central venous pressure) and closest laboratory to evaluation (lactate, venous oxygen saturation (ScVO2), arterial partial pressure of oxygen (PaO2), arterial partial pressure of carbon dioxide (PaCO2), pH, base excess (BE), bicarbonate (HCO3), carbon dioxide (CO2) arterio-venous difference, )

* Superior vena cava evaluation, Respiratory variation observed in M mode and measured. Registry of expiratory and inspiratory diameter (evaluated in the same cardiac cycle phase)
* Using Apical 5 chamber view, basal LVOT-VTI would be obtained, 3 measurements in regular rhythms and 5 measurements in irregular rhythms such as atrial fibrillation. 100 ml will be infused without changing the view and end-expiratory LVOT-VTI would be obtained a minute after infusion in the same fashion as before.
* Considering ultrasound evaluation is part of standard patient care, informed consent was waived by the ethical board.
* For analysis, the proportion of variation in superior vena cava (SVC) and VTI variation would be calculated as percentage.
* All values will be registered in a google drive table and then included in microsoft excel for coding and analyzed with Stata 12.
* Fluid responsiveness will be defined as 10% increase in VTI with the "mini bolus" fluid test, considering the minimal detectable change.
* For analysis, receiver operator curve (ROC) statistic will be done in Stata 12.
* Summary variables of the population will be presented.
* For diagnostic evaluation, the tool "roctab" for receiver operating characteristic curve will be used, obtaining cut off values, sensitivity, specificity and gray area in addition to traditional area under curve (AUC). A dichotomic value for simple orientation will be selected with an ideally balanced sensitivity and specificity for general use. Linear correlation will be explored to detect a continuous relation between SVC variation and VTI increase.
* Window success will be recorded and proportion will be analysed during the months of the study to check for performance improvements that might be expected as a learning curve effect.
* Additional data might allow post hoc analysis including window feasibility in association with clinical variables and
* After the ultrasound evaluation, the result of the 100ml test will be informed to the treating physician.
* Sample size:

Considering a possible 50% loss with inadequate acoustic window, 100 evaluated patients would achieve at least 48 included to obtain AUC 0.7. (estimating 24 to be responders and 24 not responders)

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years,
* Hospitalized in the Intensive Care Unit (ICU) with length of stay under 7 days
* Under positive pressure ventilation with no inspiratory effort,
* With hemodynamic instability (defined as abnormal peripheral perfusion or increased blood lactic or vasopressor infusion of norepinephrine >0.1 ug/kg/min to achieve adequate mean arterial pressure)

Exclusion Criteria:

* Spontaneous ventilatory effort
* Lack of venous access
* Carrier of carbapenemase or clostridium difficile
* Lack of adequate superior vena cava (SVC) window (not allowing M-mode during both respiratory phases)
* Severe aortic regurgitation
* Impossibility to measure LVOT-VTI
* Extracorporeal membrane oxygenation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ventilated critically ill patients with hemodynamic instability hospitalized in the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-07 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Fluid responsiveness | 1 minute
  An increase of 10% or more in the left ventricle velocity time integral value (average of 3 in regular rhythms or 5 in irregular rhythms) measured with cardiac ultrasound in 5 chambers apical view after the infusion of 100ml bolus of intravenous crystalloid solution.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided
Probably database will be available if asked once completed.

REFERENCES:
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Reuter DA, Chappell D, Perel A. The dark sides of fluid administration in the critically ill patient. Intensive Care Med. 2018 Jul;44(7):1138-1140. doi: 10.1007/s00134-017-4989-4. Epub 2017 Nov 11. No abstract available. PMID 29128963
- [Background] Malbrain MLNG, Van Regenmortel N, Saugel B, De Tavernier B, Van Gaal PJ, Joannes-Boyau O, Teboul JL, Rice TW, Mythen M, Monnet X. Principles of fluid management and stewardship in septic shock: it is time to consider the four D's and the four phases of fluid therapy. Ann Intensive Care. 2018 May 22;8(1):66. doi: 10.1186/s13613-018-0402-x. PMID 29789983
- [Background] Acheampong A, Vincent JL. A positive fluid balance is an independent prognostic factor in patients with sepsis. Crit Care. 2015 Jun 15;19(1):251. doi: 10.1186/s13054-015-0970-1. PMID 26073560
- [Background] Cecconi M, Hofer C, Teboul JL, Pettila V, Wilkman E, Molnar Z, Della Rocca G, Aldecoa C, Artigas A, Jog S, Sander M, Spies C, Lefrant JY, De Backer D; FENICE Investigators; ESICM Trial Group. Fluid challenges in intensive care: the FENICE study: A global inception cohort study. Intensive Care Med. 2015 Sep;41(9):1529-37. doi: 10.1007/s00134-015-3850-x. Epub 2015 Jul 11. PMID 26162676
- [Background] Bednarczyk JM, Fridfinnson JA, Kumar A, Blanchard L, Rabbani R, Bell D, Funk D, Turgeon AF, Abou-Setta AM, Zarychanski R. Incorporating Dynamic Assessment of Fluid Responsiveness Into Goal-Directed Therapy: A Systematic Review and Meta-Analysis. Crit Care Med. 2017 Sep;45(9):1538-1545. doi: 10.1097/CCM.0000000000002554. PMID 28817481
- [Background] Monnet X, Marik PE, Teboul JL. Prediction of fluid responsiveness: an update. Ann Intensive Care. 2016 Dec;6(1):111. doi: 10.1186/s13613-016-0216-7. Epub 2016 Nov 17. PMID 27858374
- [Background] Vistisen ST, Juhl-Olsen P. Where are we heading with fluid responsiveness research? Curr Opin Crit Care. 2017 Aug;23(4):318-325. doi: 10.1097/MCC.0000000000000421. PMID 28537997
- [Background] Michard F. Toward Precision Hemodynamic Management. Crit Care Med. 2017 Aug;45(8):1421-1423. doi: 10.1097/CCM.0000000000002458. No abstract available. PMID 28708687
- [Background] Vignon P, Repesse X, Begot E, Leger J, Jacob C, Bouferrache K, Slama M, Prat G, Vieillard-Baron A. Comparison of Echocardiographic Indices Used to Predict Fluid Responsiveness in Ventilated Patients. Am J Respir Crit Care Med. 2017 Apr 15;195(8):1022-1032. doi: 10.1164/rccm.201604-0844OC. PMID 27653798
- [Background] Monnet X, Osman D, Ridel C, Lamia B, Richard C, Teboul JL. Predicting volume responsiveness by using the end-expiratory occlusion in mechanically ventilated intensive care unit patients. Crit Care Med. 2009 Mar;37(3):951-6. doi: 10.1097/CCM.0b013e3181968fe1. PMID 19237902
- [Background] Monnet X, Marik P, Teboul JL. Passive leg raising for predicting fluid responsiveness: a systematic review and meta-analysis. Intensive Care Med. 2016 Dec;42(12):1935-1947. doi: 10.1007/s00134-015-4134-1. Epub 2016 Jan 29. PMID 26825952
- [Background] Biais M, Ehrmann S, Mari A, Conte B, Mahjoub Y, Desebbe O, Pottecher J, Lakhal K, Benzekri-Lefevre D, Molinari N, Boulain T, Lefrant JY, Muller L; AzuRea Group. Clinical relevance of pulse pressure variations for predicting fluid responsiveness in mechanically ventilated intensive care unit patients: the grey zone approach. Crit Care. 2014 Nov 4;18(6):587. doi: 10.1186/s13054-014-0587-9. PMID 25658489
- [Background] Muller L, Toumi M, Bousquet PJ, Riu-Poulenc B, Louart G, Candela D, Zoric L, Suehs C, de La Coussaye JE, Molinari N, Lefrant JY; AzuRea Group. An increase in aortic blood flow after an infusion of 100 ml colloid over 1 minute can predict fluid responsiveness: the mini-fluid challenge study. Anesthesiology. 2011 Sep;115(3):541-7. doi: 10.1097/ALN.0b013e318229a500. PMID 21792056
- [Background] Wu Y, Zhou S, Zhou Z, Liu B. A 10-second fluid challenge guided by transthoracic echocardiography can predict fluid responsiveness. Crit Care. 2014 May 27;18(3):R108. doi: 10.1186/cc13891. PMID 24886990
- [Background] Vieillard-Baron A, Naeije R, Haddad F, Bogaard HJ, Bull TM, Fletcher N, Lahm T, Magder S, Orde S, Schmidt G, Pinsky MR. Diagnostic workup, etiologies and management of acute right ventricle failure : A state-of-the-art paper. Intensive Care Med. 2018 Jun;44(6):774-790. doi: 10.1007/s00134-018-5172-2. Epub 2018 May 9. PMID 29744563
- [Background] Jardin F, Dubourg O, Margairaz A, Bourdarias JP. Inspiratory impairment in right ventricular performance during acute asthma. Chest. 1987 Nov;92(5):789-95. doi: 10.1378/chest.92.5.789. PMID 3665592
- [Background] Jardin F, Dubourg O, Bourdarias JP. Echocardiographic pattern of acute cor pulmonale. Chest. 1997 Jan;111(1):209-17. doi: 10.1378/chest.111.1.209. No abstract available. PMID 8996019
- [Background] Ugalde D, Haruel PA, Godement M, Prigent A, Vieillard-Baron A. Transthoracic echocardiography to evaluate the superior vena cava in critically ill patients: window description and pilot study. Intensive Care Med. 2019 Jul;45(7):1052-1054. doi: 10.1007/s00134-019-05621-1. Epub 2019 Apr 25. No abstract available. PMID 31041478
- [Background] Messina A, Dell'Anna A, Baggiani M, Torrini F, Maresca GM, Bennett V, Saderi L, Sotgiu G, Antonelli M, Cecconi M. Functional hemodynamic tests: a systematic review and a metanalysis on the reliability of the end-expiratory occlusion test and of the mini-fluid challenge in predicting fluid responsiveness. Crit Care. 2019 Jul 29;23(1):264. doi: 10.1186/s13054-019-2545-z. PMID 31358025
- [Background] Jozwiak M, Mercado P, Teboul JL, Benmalek A, Gimenez J, Depret F, Richard C, Monnet X. What is the lowest change in cardiac output that transthoracic echocardiography can detect? Crit Care. 2019 Apr 11;23(1):116. doi: 10.1186/s13054-019-2413-x. PMID 30971307
- [Derived] Ugalde D, Montoya J, Medel JN, Eisen D, Vieillard-Baron A. Diagnostic accuracy of superior vena cava variability by transthoracic echocardiography as a fluid responsiveness predictor in critically ill patients. J Crit Care. 2026 Apr;92:155420. doi: 10.1016/j.jcrc.2025.155420. Epub 2025 Dec 23. PMID 41443025